CLINICAL TRIAL: NCT03793257
Title: The EXCEL Registry: A Comprehensive Binational Registry on the Treatment and Outcomes of Patients Requiring ECMO
Brief Title: The EXCEL Registry of Patients Requiring ECMO
Status: Recruiting | Type: Observational
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Extracorporeal Life Support Organization (Unknown); National Heart Foundation, Australia (Other); The Alfred (Other); Barwon Health (Other Government); Fiona Stanley Hospital (Other); The Prince Charles Hospital (Other Government); Royal Prince Alfred Hospital, Sydney, Australia (Other); St Vincent's Hospital, Sydney (Other)
Responsible Party: Sponsor
Other Study IDs: ANZIC-RC/CH003
Record Dates: First submitted 2018-12-17; First posted 2019-01-04 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Critically Ill; Acute Respiratory Failure; Acute Heart Failure; Cardiac Arrest
Keywords: Intensive Care; Critical Care; Extracorporeal Membrane Oxygenation; Extracorporeal Life Support
MeSH Terms: conditions — Critical Illness; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ECMO is associated with significant costs, risks and requires specialist training and expertise. EXCEL is a novel, high-quality, detailed prospective registry of patients requiring ECMO in Australia and New Zealand. The registry provides information on patient selection, complications, costs and patient reported outcome measures. EXCEL uses the Theoretical Domains Framework to identify evidence-practice gaps and explore barriers and enablers to tailor implementation of evidence

DETAILED DESCRIPTION:
The aim of EXCEL is to generate a bi-national multidisciplinary network of integrated care for patients suffering acute cardiac or respiratory failure or cardiac arrest requiring extracorporeal membrane oxygenation (ECMO) to monitor long term outcomes and identify best practice.

Each year around 130,000 Australians and New Zealanders are admitted to an intensive care unit (ICU). The sickest patients in the ICU who have severe failure of the heart or lungs may require an external machine to oxygenate their blood in addition to a mechanical ventilator. This intervention, called extracorporeal membrane oxygenation (ECMO), involves circulating all of the patient's blood through large cannulae to external machinery every minute. It has the capability of completely replacing a non-functioning heart or lungs for days to weeks on end. These critically ill patients who require ECMO are the sickest in the hospital with only 42% hospital survival. The use of ECMO has doubled in Australia and New Zealand and globally over five years, and in the USA has increased by 433%.

The use of ECMO is associated with significant costs and risks, and it requires specialist training and expertise. In order to prepare for the organisation of these complex interventions in the ICU across regions, the investigators need to have accurate data on patients undergoing ECMO. The investigators monitor and review current practice in ECMO services by providing robust binational registry data to service providers and clinicians with a closed-loop feedback system. EXCEL explores barriers and enablers to evidence-based care in ECMO services and providing a platform to embed clinical trials. The investigators will translate findings with greater capacity, reach, and impact to drive measureable change in practice and improve patient-centred outcomes.

The EXCEL Partnership represents a novel, coordinated effort to create a high-quality, detailed, prospective registry of patients requiring ECMO at ECMO centres. A tailored, detailed ECMO registry (EXCEL) can be used to address specific safety concerns, clinical questions and process of care issues. As a result, EXCEL can be designed and implemented to answer new investigator-initiated, hypothesis-driven clinical questions.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to adult hospitals and receive ECMO in Australia and New Zealand

Nil Exclusion Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to hospitals with a primary diagnosis of acute heart failure, respiratory failure or cardiac arrest and received ECMO at participating ECMO centres.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Disability-free survival at 6 months, defined as alive and free of disability, measured with the World Health Organisation's Disability Assessment Schedule (WHODAS 2.0) score of <25%. | At 6 months from study enrolment
  WHODAS 2.0 measured using a trained, blinded assessor via telephone interview. The WHODAS scores are calculated using the sum of the six domain scores. These domain scores are then converted to a metric score ranging from 0 to 100 (where 0= no disability; 100= full disability)

SECONDARY OUTCOMES:
Number of participants with adverse events including major bleeding up to 28 days after ECMO, infection, thrombosis (in the ECMO cannulae or in the patient) and limb ischaemia | Up to 28 days after ECMO initiation
  All adverse events are recorded determined by treating clinician
Healthcare utilization - caseload per centre | Up to 12 months from study enrolment
  ECMO patient numbers (caseload per centre)
Healthcare utilization - ECMO initiation timing | Up to 12 months from study enrolment
  Timing of ECMO initiation by staff including an ECMO retrieval team
Healthcare utilization - number of staff members required to manage ECMO | Up to 12 months from study enrolment
  Staff numbers required for the provision of ECMO in ICU and the training required for these staff members to perform their role.
Healthcare utilization - hospital length of stay | Up to 12 months from study enrolment
  Hospital and in-patient rehabilitation length of stay including hospital readmissions and time spent in ICU
Healthcare costs | Measured from ECMO commencement to hospital discharge until 6 months following hopsital admission.
  Number of resources including staff and, equipment and blood products utilised whilst the patient was receiving hospital care until 6 months following hospital admission.
Health-related quality of life at baseline, 6 and 12 months using the EQ5D-5L | At 6 and 12 months from study enrolment. Retrospective baseline measured at 6 months.
  Measured using the EQ5D-5L, delivered by a trained, blinded assessor via telephone interview. The EQ5D includes an analogue scale that asks the patient to rate their health on a scale of 0 to 100. (Where 0= worst health imaginable; 100= best health imaginable)
Number of patients with disability at 6 and 12 months | At 6 and 12 months from study enrolment
  Measured using the WHODAS 2.0, delivered by a trained, blinded assessor via telephone interview
Psychological function at 12 months | At 12 months from study enrolment
  Measured using the EQ5D-5L, delivered by a trained, blinded assessor via telephone interview
Return to work at 6 months | At 6 months from study enrolment
  Return to work measured bu the WHODAS 2.0, delivered by a trained, blinded assessor via telephone interview
Disability at baseline, 6 and 12 months | Measured at 6 and 12 months. Retrospective baseline disability measured at 6 months.
  Patient reported disability using a disability scale, delivered by a trained, blinded assessor via telephone interview
Activities of daily living at 6 and 12 months | Measured at 6 and 12 months
  Activities of daily living measured at 6 and 12 month using the ADL and IADL, delivered by a trained, blinded assessor via telephone interview
Cognitive function at 12 months | Measured at 12 months
  Cognitive function measured at 12 months using the MOCA Blind, delivered by a trained, blinded assessor via telephone interview
Number patients who survive to 12 months following ECMO initiation | At 12 months from study enrolment
  Measured by Research Coordinators at each of the participating sites

CONTACTS AND LOCATIONS:
Overall Officials: Carol L Hodgson, PhD, Study Chair — Australian and New Zealand Intensive Care Research Centre
Locations (29):
- Australia (28):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, Newcastle, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - St George Hospital, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Prince Charles Hospital, Chermside, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Sunshine Coast University Hospital, Sunshine Coast, Queensland
  - Townsville Hospital, Townsville, Queensland
  - Royal Adelaide Hosptial, Adelaide, South Australia
  - Flinders Medical Centre, Adelaide, South Australia
  - Launceston General Hospital, Launceston, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - University Hospital Geelong, Geelong, Victoria
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - St Vincent's Hospital Melbourne, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Epworth Hospital, Richmond, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Fiona Stanley Hospital, Perth, Western Australia
- Auckland City hospital, Auckland, New Zealand

REFERENCES:
- [Result] Hodgson CL, Higgins AM, Bailey MJ, Anderson S, Bernard S, Fulcher BJ, Koe D, Linke NJ, Board JV, Brodie D, Buhr H, Burrell AJC, Cooper DJ, Fan E, Fraser JF, Gattas DJ, Hopper IK, Huckson S, Litton E, McGuinness SP, Nair P, Orford N, Parke RL, Pellegrino VA, Pilcher DV, Sheldrake J, Reddi BAJ, Stub D, Trapani TV, Udy AA, Serpa Neto A; EXCEL Study Investigators on behalf of the International ECMO Network and the Australian and New Zealand Intensive Care Society Clinical Trials Group. Incidence of death or disability at 6 months after extracorporeal membrane oxygenation in Australia: a prospective, multicentre, registry-embedded cohort study. Lancet Respir Med. 2022 Nov;10(11):1038-1048. doi: 10.1016/S2213-2600(22)00248-X. Epub 2022 Sep 26. PMID 36174613
- [Result] Fulcher BJ, Nicholson AJ, Linke NJ, Berkovic D, Hodgson CL; EXCEL Study Investigators and the International ECMO Network. The perceived barriers and facilitators to implementation of ECMO services in acute hospitals. Intensive Care Med. 2020 Nov;46(11):2115-2117. doi: 10.1007/s00134-020-06187-z. Epub 2020 Jul 23. No abstract available. PMID 32705292
- [Result] Linke NJ, Fulcher BJ, Engeler DM, Anderson S, Bailey MJ, Bernard S, Board JV, Brodie D, Buhr H, Burrell AJC, Cooper DJ, Fan E, Fraser JF, Gattas DJ, Higgins AM, Hopper IK, Huckson S, Litton E, McGuinness SP, Nair P, Orford N, Parke RL, Pellegrino VA, Pilcher DV, Sheldrake J, Reddi BAJ, Stub D, Trapani TV, Udy AA, Hodgson CL; EXCEL Investigators. A survey of extracorporeal membrane oxygenation practice in 23 Australian adult intensive care units. Crit Care Resusc. 2020 Jun;22(2):166-170. doi: 10.51893/2020.2.sur7. No abstract available. PMID 32389109
- [Derived] Brown A, Dennis M, Rattan N, Nanjayya V, Burrell A, Serpa Neto A, Hodgson C; EXCEL (a Comprehensive Binational Registry on the Treatment and Outcomes of Patients Requiring Extracorporeal Membrane Oxygenation [ECMO]) Study Investigators and the International ECMO Network. Neurologic Complications During Venoarterial Extracorporeal Membrane Oxygenation and Their Implications for 6-Month Patient-Centered Outcomes. Crit Care Med. 2026 Jan 1;54(1):175-186. doi: 10.1097/CCM.0000000000006938. Epub 2025 Nov 10. PMID 41212045
- [Derived] Serpa Neto A, Higgins AM, Bailey MJ, Anderson S, Bernard S, Fulcher BJ, Jones A, Linke NJ, Board JV, Brodie D, Buhr H, Burrell AJC, Cooper DJ, Fan E, Fraser JF, Gattas DJ, Hopper IK, Huckson S, Litton E, McGuinness SP, Nair P, Orford N, Parke RL, Pellegrino VA, Pilcher DV, Dicker C, Reddi BAJ, Stub D, Trapani TV, Udy AA, Hodgson CL; EXCEL Study Investigators on behalf of the International ECMO Network (ECMONet). Long-Term Functional Outcomes in the First 12 Months After VA-ECMO in Adult Patients: A Prospective, Multicenter Study. Circ Heart Fail. 2025 Jun;18(6):e012476. doi: 10.1161/CIRCHEARTFAILURE.124.012476. Epub 2025 Apr 29. PMID 40298907
- See also: EXCEL Registry Website — https://www.monash.edu/medicine/sphpm/excel/home